CLINICAL TRIAL: NCT05141292
Title: A Registry Study of Biomarkers in Mitral Valve Disease
Brief Title: A Registry Study of Biomarkers in Mitral Valve Disease (BIOMS-MVD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BIOMS-MVD
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The registry study aims to discover the prognostic value of bio-markers in mitral valve disease

DETAILED DESCRIPTION:
The purpose of this study is to investigate the prognostic value of biomarkers in mitral valve disease.Patients with confirmed diagnosis of mitral valve disease are enrolled.The primary outcome is all-cause mortality based on the death certificates. The secondary outcome is readmission for heart failure and all-cause mortality/readmission for heart failure according to the patients' medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed with mitral valve disease in Beijing Anzhen Hospital from April 2016 to December 2019
* The operator performs more than 25 mitral valve operations per year / the operator unit has surgeons who complete 50 operations per year

Exclusion Criteria:

* Age ≤ 18 years
* Failure to obtain medical records and ultrasound data
* Refuse follow-up

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure accorrding to Inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of death (all cause) | 1 years of follow-up
  Number of death within 2 years of discharge

SECONDARY OUTCOMES:
Number of rehospitalizations | 1 years of follow-up
  Number of heart failure related hospitalization within 1 years of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jie Du, Study Director — The Key Laboratory of Remodeling-Related Cardiovascular Disease, Ministry of Education, Beijing Anzhen Hospital, Capital Medical University, Beijing Institute of Heart,Lung and Blood Vessel Diseases
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhou N, Zhang K, Qiao B, Chen C, Guo X, Fu W, Zheng J, Du J, Dong R. Personalized risk prediction of mortality and rehospitalization for heart failure in patients undergoing mitral valve repair surgery. Front Cardiovasc Med. 2024 Nov 1;11:1470987. doi: 10.3389/fcvm.2024.1470987. eCollection 2024. PMID 39553845
- [Derived] Zhou N, Ji Z, Li F, Qiao B, Lin R, Jiang W, Zhu Y, Lin Y, Zhang K, Li S, You B, Gao P, Dong R, Wang Y, Du J. Machine Learning-Based Personalized Risk Prediction Model for Mortality of Patients Undergoing Mitral Valve Surgery: The PRIME Score. Front Cardiovasc Med. 2022 Apr 1;9:866257. doi: 10.3389/fcvm.2022.866257. eCollection 2022. PMID 35433879